CLINICAL TRIAL: NCT04476693
Title: Metabolic Responses to Breakfast Consumption Versus Omission in Adolescent Girls
Brief Title: Metabolic Responses to Breakfast in Adolescent Girls
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bedfordshire (Other)
Collaborators: British Nutrition Foundation (Unknown)
Responsible Party: Principal Investigator, Dr Rebecca Jones, Lecturer in Exercise Physiology, University of Bedfordshire
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: UBedfordshire
Record Dates: First submitted 2020-07-09; First posted 2020-07-20 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Postprandial Hyperglycemia
Keywords: cardiovascular disease; diabetes
MeSH Terms: conditions — Hyperglycemia; Cardiovascular Diseases; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Two experimental trials will be completed in a randomised counterbalanced order: BC and BO. A standardised lunch will be provided three hours after breakfast consumption (BC) or after water consumption during breakfast omission (BO). Finger prick blood samples for the analysis of plasma glucose, insulin and triaclglycerol and expired gas samples for the analysis of substrate oxidation will be taken throughout the trials. An incremental cycling exercise test with 4 minute stages will be performed 2 h after lunch for the determination of maximum fat oxidation (MFO) and intensity at which MFO occurred (i.e., Fatmax). The OMNI scale will be used to evaluate the perceived exertion at the end of each cycling stage. PA enjoyment will be evaluated using Physical Activity Enjoyment Scale (PACES).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breakfast Consumption (BC) (Experimental): The consumption of a standardised breakfast followed by a standardised lunch 3-h after the last mouthful of breakfast meal. All the ingredients of the breakfast and lunch provided will be weighed, with the portion sizes calculated based on individual resting metabolic rate (RMR). The participants were instructed to consume the meals provided within 15 min. A minimum of seven days washout period will be provided to avoid carry-over effects between conditions.
  The standardised lunch will consist of white bread without crust (Tesco), margarine 'Butter Me Up Spread' (Tesco), strawberry jam (Tesco), salted crisps (Walkers) and sparkling glucose drink (Lucozade Energy Original). This carbohydrate-rich high glycameic index lunch was designed to trigger quick and exaggerated glucose and insulin response.
  Interventions: Other: Breakfast consumption
- Breakfast omission (BO) (Experimental): Participant will consume water, the individual volume of which was calculated based on the liquid content of the breakfast. A standardised lunch will be consumed 3-h after the last mouthful of water. All the ingredients of the breakfast and lunch provided were weighed, with the portion sizes calculated based on individual resting metabolic rate (RMR). The participants were instructed to consume the meals provided within 15 min. A minimum of seven days washout period was provided to avoid carry-over effects between conditions.
  The standardised lunch consists of white bread without crust (Tesco), margarine 'Butter Me Up Spread' (Tesco), strawberry jam (Tesco), salted crisps (Walkers) and sparkling glucose drink (Lucozade Energy Original). This carbohydrate-rich high glycameic index lunch was designed to trigger quick and exaggerated glucose and insulin response.
  Interventions: Other: Breakfast Omission

INTERVENTIONS:
Other: Breakfast consumption — Consumption of breakfast: The breakfast provided was designed based on the "characteristics of an ideal breakfast" outlined in Giovannini et al., (2008). The breakfast provided in the present study will include the following: all-bran cereals (Kellogg's), semi-skimmed milk (Tesco), Royal Gala Apple (Tesco) and Orange Juice from Concentrate (Tesco) containing the amount of carbohydrates usually consumed at breakfast in the UK (Reeves et al., 2013). The portion for each participant will contain 0.06 g of carbohydrate per kcal of measured RMR. As the portion size (20% of daily calorie intake) will be calculated based on individual RMR , no leftovers will be allowed.
  Arms: Breakfast Consumption (BC)
Other: Breakfast Omission — Omission of breakfast. Participants will consume water within 15 min, the individual volume of which will be calculated based on the liquid content of the breakfast [milk (ml)+ orange juice (ml)].
  Arms: Breakfast omission (BO)

SUMMARY:
Breakfast consumption (BC) is frequently associated with a healthy lifestyle, healthy body weight and favourable cardiometabolic health. Research from studies in adults suggests that breakfast skipping causes elevated plasma glucose and insulin concentrations after lunch. However, there is currently no evidence to suggest a similar metabolic response in adolescent girls, a population that frequently skips breakfast. The primary purpose of this study is to examine the effects of BC versus breakfast omission (BO) on metabolic responses after lunch in healthy adolescent girls.

DETAILED DESCRIPTION:
Breakfast consumption (BC) is habitually associated with a healthy lifestyle (e.g., diet and physical activity), reduced adiposity and favourable cardiometabolic health profiles in children, adolescents and adults. Experimental research in adults has shown that breakfast consumption reduces the glycaemic and insulinemic response to lunch when compared with breakfast omission; this has been termed 'the second meal effect'. Further, breakfast consumption may improve exercise performance and increase free-living physical activity energy expenditure in adults. Understanding the postprandial metabolic responses to BC and breakfast omission (BO) in adolescent girls is particularly important, as this population frequently skips breakfast and have low physical activity levels. Yet, adolescent girls may respond differently to adults due to their distinct metabolic profiles, and past research has not targeted this population. The primary aim of this research is to examine whether BC versus BO affects postprandial glycaemic and insulinemic responses to lunch in adolescent girls. Secondly, it aims to examine the lipaemic and substrate oxidation responses during rest, substrate oxidation during an exercise bout performed later in the day, and physical activity enjoyment during the exercise bout.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 11 to 14 years old
2. Female
3. Healthy weight Body Mass Index centile (between the 3rd and 91st centile - Cole et al 2000)

Exclusion Criteria:

1. Allergies to the breakfast and lunch ingredients
2. Fitted with a pacemaker
3. Unable to walk
4. Health related issues that could be affected by participation in the study (e.g., uncontrolled exercise-induced asthma, diabetes, epilepsy)

Ages: 11 Years to 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Post-lunch area under the curve (AUC) for glucose. | 2 hours
  Net incremental AUC and total AUC for 2-hour period post lunch in each condition will be calculated for plasma glucose. Five finger prick blood samples will be taken at 15, 30, 60, 90 and 120 minutes post lunch.
Total trial area under the curve (AUC) for glucose. | 5 hours
  Net incremental AUC and total AUC for the 5-hour entire trial period in each condition will be calculated for plasma glucose. Finger prick blood samples will be taken at at 0 (baseline), 30, 60, 120 and 180 min after breakfast consumption or omission and at 15, 30, 60, 90 and 120 minutes after lunch consumption.
Post-lunch area under the curve (AUC) for insulin. | 2 hours
  Net incremental AUC and totral AUC for 2-hour period post lunch in each condition will be calculated for plasma insulin. Five finger prick blood samples will be taken at 15, 30, 60, 90 and 120 minutes post lunch.
Total trial area under the curve (AUC) for insulin. | 5 hours
  Net incremental AUC and total AUC for the 5-hour entire trial period in each condition will be calculated for plasma insulin. Finger prick blood samples will be taken at at 0 (baseline), 30, 60, 120 and 180 min after breakfast consumption or omission and at 15, 30, 60, 90 and 120 minutes after lunch consumption.

SECONDARY OUTCOMES:
Post-lunch resting substrate oxidation | 2 hours
  Substrate oxidation (fat and carbohydrate) rates will be estimated using indirect calorimetry from expired air samples at four time points following lunch (30, 60, 90 and 120 minutes).
Total trial resting substrate oxidation. | 5 hours
  Substrate oxidation (fat and carbohydrate) rates will be estimated using indirect calorimetry from expired air samples at baseline and at 4 time points after breakfast (30, 60, 120 and 180 minutes) and 4 time points following lunch (30, 60, 90 and 120 minutes).
Maximum fat oxidation rate during exercise | During exercise (approximately 30 minutes)
  An incremental 7-stage cycling test will be performed 2 hours after lunch for the determination of maximum fat oxidation. Each stage will last 4 minutes in duration, where participants will keep a steady pedalling rate of 60 revolutions per minute. The intensity for each stage was calculated based on the percentage (0%, 20%, 30%, 40%, 50%, 60%, 70%) of the theoretical maximal aerobic power. Fat oxidation rates will be estimated during the final minute of each stage using indirect calorimetry.
Fatmax during exercise | During exercise (approximately 30 minutes)
  An incremental 7-stage cycling test will be performed 2 hours after lunch for the determination of maximum fat oxidation. Each stage will last 4 minutes in duration, where participants will keep a steady pedalling rate of 60 revolutions per minute. The intensity for each stage was calculated based on the percentage (0%, 20%, 30%, 40%, 50%, 60%, 70%) of the theoretical maximal aerobic power. Fat oxidation rates will be estimated during the final minute of each stage using indirect calorimetry. The intensity at which maximum fat oxidation occurs will be defined as Fatmax.
Physical activity enjoyment | Following exercise (approximately 5-10 minutes post)
  Physical activity enjoyment measured using Physical Activity Enjoyment Scale (PACES) during the Fatmax incremental exercise test. The scale is composed of 16 statements (9 positive and 7 negative) which begin with the phrase "When I am physically active…". The participants must answer by giving an answer from 1 "disagree a lot" to 5 "agree a lot" to each statement. The average score of the positive statements is calculated to be used in the analysis.
Post-lunch area under the curve (AUC) for triaclyglycerol | 2 hour
  Net incremental AUC and total AUC for the 2-hour period post lunch in each condition will be calculated for plasma triaclyglycerol. Five finger prick blood samples will be taken at 15, 30, 60, 90 and 120 minutes post lunch.
Total trial area under the curve (AUC) for triaclyglycerol | 5 hours
  Net incremental AUC and total AUC for the 5-hour entire trial period in each condition will be calculated for plasma triacylglycerol. Finger prick blood samples will be taken at at 0 (baseline), 30, 60, 120 and 180 min after breakfast consumption or omission and at 15, 30, 60, 90 and 120 minutes after lunch consumption.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Bedfordshire, Bedford, Bedfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No